CLINICAL TRIAL: NCT04806646
Title: A Phase II, Open-label Study Improving Compliance and Time of Treatment After Obtaining Complete Response Through a Tailored Schedule of Sonidegib in Locally Advanced Basal Cell Carcinomas (BCC) - the SONIBEC Trial
Brief Title: Tailored Sonidegib Schedule After Complete Response in BCC
Acronym: SONIBEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SONIBEC
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Locally Advanced Basal Cell Carcinoma
MeSH Terms: interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Treatment (Experimental): One cycle of therapy is defined as 28 days of sonidegib. The patient will start with TS1 schedule.
  * TS1: assumption 14 days on and 14 days off. TS1 may be temporary interrupted for any grade 2 or 3 toxicity (excluding alopecia) until return to grade 1. If the patient experiences any grade 3 or 2 side effects lasting for more than 28 days, at treatment resumption they will start the TS2 schedule.
  * TS2: assumption 7 days on and 21 days off. TS2 may be temporary interrupted for any grade 2 or 3 toxicity (excluding alopecia) until return to grade 1. If the patient experiences any grade 3 or 2 side effects lasting for more than 28 days, he/she is discontinued from the study.
  If progression of disease is observed (during TS1 or TS2) the patient is discontinued from the study.
  Interventions: Drug: Sonidegib

INTERVENTIONS:
Drug: Sonidegib — TS1: assumption 14 days on and 14 days off. TS2: assumption 7 days on and 21 days off.
  Other Names: Odomzo

SUMMARY:
Adult patients with locally advanced BCC, not amenable to surgical treatment and who obtained a complete response (CR) to Hedgehog inhibitors are administered a tailored schedule of the study drug. The tailored schedule consists of a change in the time of drug assumption. It implements some weeks of assumption and some weeks of suspension of sonidegib rather than a continuous administration.

DETAILED DESCRIPTION:
One cycle of therapy is defined as 28 days of sonidegib. The patient will start with first schedule.

* Treatment schedule 1 (TS1): assumption 14 days on and 14 days off. TS1 may be temporary interrupted for any grade 2 or 3 toxicity (excluding alopecia) until return to grade 1. If the patient experiences any grade 3 or 2 side effects lasting for more than 28 days, at treatment resumption they will start the TS2 schedule.
* Treatment schedule 2 (TS2): assumption 7 days on and 21 days off. TS2 may be temporary interrupted for any grade 2 or 3 toxicity (excluding alopecia) until return to grade 1. If the patient experiences any grade 3 or 2 side effects lasting for more than 28 days, he/she is discontinued from the study.

If progression of disease is observed (during TS1 or TS2) the patient is discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed informed consent, including consent to photographs of lesions.
2. Age ≥ 18 years.
3. Histologic confirmation of locally advanced BCC lesion.
4. Patients with BCCs already in treatment with Hedgehog inhibitor sonidegib for:

   * BCC that has recurred in the same location after three or more surgical procedures and/or curative resection is deemed unlikely
   * multifocal BCC or extensive tumours with bleeding or infected areas
   * anticipated substantial morbidity and/or deformity from surgery (e.g. removal of all or part of a facial structure, such as nose, ear, eyelid, eye; or requirement for limb amputation)
   * multiple BCCs not amenable to surgical treatment because of oncologic or clinical reasons
5. Patient having shown a complete response (CR) to Hedgehog inhibitor sonidegib within the 3 months prior to the screening. In BCC every effort should be made to obtain histologic confirmation of CR mainly in case of doubt, performing several biopsies in the sites where disease was present. CR must have been confirmed by 2 consecutive radiologic exams and by visual and dermoscopic examinations.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Adequate hematopoietic capacity, defined as the following:

   * Haemoglobin > 8.5 g/dl
   * Absolute neutrophil count (ANC) ≥ 1000/mmc
   * Platelet count ≥ 75,000/mmc
8. Adequate hepatic and renal function, defined as the following:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN), Total bilirubin ≤ 1.5 × ULN or within 3 × ULN for patients with documented Gilbert syndrome
   * Calculated serum creatinine clearance (CrCl) ≥ 30 mL/min
9. For women of childbearing potential, a negative pregnancy test within 7 days prior to commencement of dosing is required
10. Women of child-bearing potential must use two methods of acceptable contraception including one highly effective method and a barrier method, as directed by their physician, during treatment and for at least 20 months after completion of study treatment. Highly effective methods of contraception are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (e.g., implants, injectables, combined oral contraception, or intra-uterine devices). Check Appendix B for details.
11. Participant must agree to not breastfeed during the study and for 20 months after the last dose of study treatment.
12. For male patients with female partners of childbearing potential, agreement to use a condom, even after a vasectomy, during sexual intercourse with female partners while being treated with sonidegib, and for 6 months after the last dose was received.
13. Agreement not to donate blood or blood products during the study and for at least 20 months after the last dose was received.
14. For male patients, agreement not to donate sperm during treatment and for 6 months after the last dose was received.

Exclusion Criteria:

1. Metastatic BCC.
2. Inability or unwillingness to swallow capsules.
3. Inability or unwillingness to comply with study procedures.
4. Pregnancy or lactation.
5. Concurrent non-protocol-specified anti-tumour therapy (e.g., chemotherapy, other targeted therapy, radiation therapy, or photodynamic therapy, including participation in an experimental drug study).
6. Uncontrolled medical illness, including advanced malignancies, at the discretion of the Investigator.
7. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk for treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2024-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Maintaining tailored treatment | 12 months
  Proportion of patients maintaining the tailored treatment with sonidegib 12 months after enrolment into the study.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, MD, Principal Investigator — Gono - ASST Spedali Civili Brescia
Locations (1):
- Asst Degli Spedali Civili Di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No